CLINICAL TRIAL: NCT06187376
Title: Evaluating the Safety and Acceptability of Using Chinese Herbal Medicine in Patients With Primary Dysmenorrhea: A Randomized-controlled Trial
Brief Title: Chinese Herbal Medicine for Gynecologic Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn due to inability to determine path forward regarding study design between sponsor and institutional staff.
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: Zenchi, Inc. (Industry)
Responsible Party: Principal Investigator, Jenny Tang, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-23-01101
Record Dates: First submitted 2023-12-13; First posted 2024-01-02 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Dysmenorrhea
MeSH Terms: conditions — Dysmenorrhea | interventions — Rab geranylgeranyltransferase

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chinese Herbal Medicine (CHM) herbal tincture (Experimental): Chinese herbal tincture
  Interventions: Drug: Chinese Herbal Medicine (CHM) supplement
- Placebo (Placebo Comparator): Matching placebo tincture.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Chinese Herbal Medicine (CHM) supplement — Dropper of tincture by mouth for 12 weeks.
  Arms: Chinese Herbal Medicine (CHM) herbal tincture
Drug: Placebo — Matching placebo tincture.
  Arms: Placebo

SUMMARY:
This is a prospective randomized-controlled trial looking at the safety and acceptability of using Chinese herbal medicine in patients with primary dysmenorrhea. The research team hopes to enroll 100 patients, 50 of whom will be randomized to receive the herbal tincture and 50 who will receive a placebo tincture. Patients will be enrolled and using the assigned tincture for twelve weeks. The research team will assess safety as a primary outcome by the presence or absence of adverse events related to study protocol during the period of participation.

ELIGIBILITY:
Inclusion Criteria:

* Female aged 18-36 are met:
* Self-reported pain or discomfort during menstruation, as indicated by Grade 1 or higher on the verbal multidimensional scoring system
* May experience regular menstrual cycle and period must be <7 days in duration
* May be on birth control
* Must know or can estimate the date of the next cycle/period
* May find blood clots in menstrual blood
* Must be in good health (doesn't report any medical conditions asked in the screening questionnaire)
* Following a stable, consistent diet regimen
* Follow a stable, consistent exercise regimen and are willing, for the duration of the study, to not decrease or increase the amount of exercise in their regimen
* Agree to refrain from any lifestyle changes that may affect their menstrual cycle for the duration of the study (for example, getting on or off hormonal birth control, reducing the amount of exercise)
* Follow a stable consistent regimen when using any other interventions, such as massage, chiropractic medicine, or acupuncture; agree not to increase or decrease the number of their other interventions
* Willingness to adhere to the dietary supplement regimen
* Willingness to refrain from any other dietary supplements targeting the menstrual cycle during the study period
* Is able to communicate in English
* Is willing and able to share feedback via REDCap
* Must provide written informed consent (ICF)

Exclusion Criteria:

* Do not experience a menstrual cycle
* Cannot estimate the onset of their next menstrual cycle
* Do not experience menstrual pain or cramping
* Follow an extreme diet intervention
* Experienced severe weight loss in the past 3 months prior to study participation
* If currently taking allowed supplements, the dosage needs to remain the same throughout the entirety of the study
* Food intolerances/allergies that require an EpiPen
* Known allergic reaction to any of the test product ingredients
* Currently pregnant, want to become pregnant for the duration of the study, or who are breastfeeding
* Previous users of Elix Cycle Balance
* Having more than 3 alcoholic drinks a day
* Have been diagnosed with the following conditions: PCOS, endometriosis, PMDD, adenomyosis, Hashimoto's, anorexia, bulimia, orthorexia, binge eating, any other eating disorder
* Smokers
* Not been on a stable dose of birth control for the past 6 months

Ages: 18 Years to 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

PRIMARY OUTCOMES:
Presence or absence of any adverse events | up to 3 months
  Presence or absence of any adverse events related to the study protocol during the time of participation.

SECONDARY OUTCOMES:
Dysmenorrhea Symptom Interference (DSI) Scale | up to 3 months
  Dysmenorrhea Symptom Interference (DSI) Scale: Is a nine-item validated measure of symptoms associated with dysmenorrhea including working ability, location, intensity, and days of pain. Symptoms are ranked from 1 (not at all) to 5 (very much) with regard to their interference with various aspects of their daily function. To generate total scores, the nine-items are averaged, thus total scale scores range from 1-5, with higher scores indicating greater interference of dysmenorrhea symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Tavella, Study Director — Icahn School of Medicine
Locations (1):
- Mount Sinai Faculty Practice Associates, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  To achieve aims in the approved proposal. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in the University's data warehouse but without investigator support other than deposited metadata.